CLINICAL TRIAL: NCT03013686
Title: The Treatment of Periappendicular Abscess After the Acute Phase (PeriAPPAC): a Randomized Clinical Trial Interval Appendectomy Versus Follow-up
Brief Title: The Treatment of Periappendicular Abscess After the Acute Phase
Acronym: PeriAPPAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, Principal investigator, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PeriAPPAC
Record Dates: First submitted 2016-08-19; First posted 2017-01-06 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Periappendicular Abscess
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval Appendectomy (Active Comparator): The periappendicular abscess, diagnosed by a CT-scan or MRI, is initially treated conservatively with antibiotic therapy and with drainage, if necessary.
  Interval appendectomy is performed at two months after the primary treatment, all patients also undergo colonoscopy prior to appendectomy.
  Interventions: Procedure: Interval appendectomy
- Follow-up with MRI (Active Comparator): The periappendicular abscess, diagnosed by a CT-scan or MRI, is initially treated conservatively with antibiotic therapy and with drainage, if necessary.
  The patients undergo abdominal magnetic resonance imaging at two months after the primary treatment, all patients also undergo colonoscopy right after the MRI.
  Interventions: Procedure: Follow-up with MRI

INTERVENTIONS:
Procedure: Interval appendectomy — Laparoscopic appendectomy
  Arms: Interval Appendectomy
Procedure: Follow-up with MRI — Abdominal MRI
  Arms: Follow-up with MRI

SUMMARY:
The PeriAPPAC trial is a prospective randomised study comparing interval laparoscopic appendectomy with follow-up MRI in patients with initially successfully treated periappendicular abscess.

Periappendicular abscess is generally initially treated conservatively with antibiotic therapy and if necessary, drainage. Operative treatment in the acute abscess phase is associated with increased morbidity and thus complicated appendicitis with a periappendicular abscess is initially treated conservatively. However, there is debate on whether interval appendectomy is required.

After initial successful conservative treatment of a CT- or MRI-diagnosed periappendicular abscess, patients enrolled in the PeriAPPAC study are randomised either to interval appendectomy or to follow-up with MRI at two months after the initial treatment. All patients also undergo a colonoscopy, appendectomy patients prior to surgery and MRI patients after the MRI (outpatient visit at endoscopy unit with information on the MRI).

The primary endpoint is the treatment success in both treatment arms. In the interval appendectomy evaluated as possible morbidity related to appendectomy and in the follow-up treatment arm as possible recurrence of the appendicitis and/or abscess during a one-year follow-up.

The PeriAPPAC study is a multi centre trial and the participating hospitals are Turku University Hospital, Oulu University Hospital, Tampere University Hospital, Kuopio University Hospital and Seinäjoki Central Hospital.

DETAILED DESCRIPTION:
The PeriAPPAC trial is a prospective randomised study comparing interval laparoscopic appendectomy with follow-up MRI in patients with initially successfully treated periappendicular abscess.

Periappendicular abscess is generally initially treated conservatively with antibiotic therapy and if necessary, drainage. Operative treatment in the acute abscess phase is associated with increased morbidity and thus complicated appendicitis with a periappendicular abscess is initially treated conservatively. However, there is debate on whether interval appendectomy is required.

After initial successful conservative treatment of a CT- or MRI-diagnosed periappendicular abscess, patients enrolled in the PeriAPPAC study are randomised either to interval appendectomy or to follow-up with MRI at two months after the initial treatment. All patients also undergo a colonoscopy, appendectomy patients prior to surgery and MRI patients after the MRI (outpatient visit at endoscopy unit with information on the MRI).

The primary endpoint is the treatment success in both treatment arms. In the interval appendectomy evaluated as possible morbidity related to appendectomy and in the follow-up treatment arm as possible recurrence of the appendicitis and/or abscess during a one-year follow-up.

The PeriAPPAC study is a multi centre trial and the participating hospitals are Turku University Hospital, Oulu University Hospital, Tampere University Hospital, Kuopio University Hospital and Seinäjoki Central Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* CT- or MRI-diagnosed periappendicular abscess, that has initially undergone successful conservative treatment with antibiotic therapy and drainage, if necessary

Exclusion Criteria:

* Suspicion of a tumour on CT or MRI
* Age under 18 years or over 60 years
* Pregnancy or lactating
* Allergy to contrast media or iodine
* Renal insufficiency
* Metformin medication (DM)
* Unsuccessful initial conservative treatment of periappendicular abscess
* Lack of co-operation (unable to give consent)
* A severe medical condition
* Previous acute appendicitis treated conservatively with antibiotics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-01-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success | One year after the intervention
  Treatment success in both treatment arms. In the interval appendectomy evaluated as possible morbidity related to appendectomy and successful appendectomy and in the follow-up treatment arm as possible recurrence of the appendicitis and/or abscess during a one-year follow-up

SECONDARY OUTCOMES:
Possible appendiceal or colon tumours | 1-10 years
  The incidence of possible tumours
Possible diagnosis of Crohn's disease | 1-10 years
  The incidence of possible Crohn's disease
The length of hospital stay | up to one year
  Length of hospital stay
Sick leave | up to one year
  Sick leave (days)
Overall morbidity | Up to 10 years, time points 1, 3, 5 and 10 years
  Complications related to disease / intervention
Mortality | Up to 10 years
  Mortality
Treatment costs | Up to 10 years
  Overall treatment costs

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mallinen J, Rautio T, Gronroos J, Rantanen T, Nordstrom P, Savolainen H, Ohtonen P, Hurme S, Salminen P. Risk of Appendiceal Neoplasm in Periappendicular Abscess in Patients Treated With Interval Appendectomy vs Follow-up With Magnetic Resonance Imaging: 1-Year Outcomes of the Peri-Appendicitis Acuta Randomized Clinical Trial. JAMA Surg. 2019 Mar 1;154(3):200-207. doi: 10.1001/jamasurg.2018.4373. PMID 30484824